CLINICAL TRIAL: NCT03267186
Title: A Phase 2 Study of Ibrutinib Maintenance After Reduced-Intensity Conditioning and Allogeneic Hematopoietic Cell Transplantation for Acute Leukemia
Brief Title: Ibrutinib in Preventing Acute Leukemia in Patients After Reduced-Intensity Conditioning and Stem Cell Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Andrew Rezvani (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor-Investigator, Andrew Rezvani, Associate Professor of Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-38934; NCI-2017-00125 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB-38934 (Other: Stanford IRB); BMT302 (Other: OnCore)
Record Dates: First submitted 2017-08-28; First posted 2017-08-30 (Actual); Results first posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Acute Biphenotypic Leukemia; Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia; Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Hematopoietic Cell Transplantation Recipient
MeSH Terms: conditions — Leukemia, Biphenotypic, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Prevention (ibrutinib) (Experimental): Beginning 60-90 days after allogeneic HCT, patients receive ibrutinib PO QD for up to 18 months post-transplant in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Ibrutinib; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA-032765; Imbruvica; PCI-32765
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies how well ibrutinib works in preventing acute leukemia in patients after reduced-intensity conditioning and stem cell transplant. Ibrutinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To reduce the incidence of relapse at 18 months after reduced-intensity conditioning (RIC) and allogeneic hematopoietic cell transplantation (HCT) for acute myeloid leukemia (AML), acute lymphoblastic leukemia (ALL), and chronic myeloid leukemia (CML) in blast crisis from a historical baseline of 45% to 25%, using ibrutinib maintenance therapy.

SECONDARY OBJECTIVES:

I. To study the incidence and severity of post-transplant complications in subjects receiving ibrutinib maintenance after allogeneic HCT.

II. To study the incidence of infectious complications in subjects receiving maintenance ibrutinib after allogeneic HCT.

III. To study the impact of ibrutinib maintenance on minimal residual disease after RIC and allogeneic HCT.

IV. To study the impact of maintenance ibrutinib on immune reconstitution and alloreactivity after allogeneic HCT, specifically on Th1/ Th2 polarization, T follicular cell number, T and B cell repertoire, serum immunoglobulin levels, and alloantibody formation.

OUTLINE:

Beginning 60-90 days after allogeneic HCT, patients receive ibrutinib orally (PO) once daily (QD) for up to 18 months post-transplant in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* INCLUSION CRITERIA FOR ENROLLMENT (PRE-TRANSPLANT)
* Diagnosis of acute myeloid leukemia (AML), acute biphenotypic leukemia, or acute lymphoblastic leukemia (ALL); CML transformed to blast crisis is eligible
* Planned allogeneic HCT using fludarabine phosphate (FLU)/melphalan hydrochloride (MEL) or FLU/busulfan (BU) conditioning
* Planned graft versus host disease (GVHD) prophylaxis consisting of tacrolimus (TAC)/methotrexate (MTX) or TAC/sirolimus (SRL)
* Human leukocyte antigen (HLA) identical sibling donor, HLA matched unrelated donor, or donor mismatched at 1 HLA allele or antigen
* Less than or equal to 5% blasts on bone marrow examination within 60 days of starting conditioning
* Age >= 18 years and =< 70 years
* Able to give informed consent
* Subjects will be eligible if their planned conditioning regimen for allogeneic HCT consists of one of the two following standard reduced intensity conditioning regimens:

  * FLU/MEL: fludarabine phosphate (fludarabine) 120 to 180 mg/m^2; melphalan hydrochloride (melphalan) =< 150 mg/m^2
  * FLU/BU: fludarabine 120 to 180 mg/m^2; busulfan =< 8 mg/kg orally or =< 6.4 mg/kg intravenously
* Subjects will be eligible if their planned post grafting immunosuppression consists of one of the two following regimens:

  * TAC/MTX: tacrolimus (oral or intravenous) and intravenous methotrexate administered according to institutional standard practice.
  * TAC/SRL: tacrolimus (oral or intravenous) and oral sirolimus, administered according to institutional standards of care
* INCLUSION CRITERIA (PRIOR TO IBRUTINIB ADMINISTRATION)
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Absolute neutrophil count (ANC) > 0.75 x 10^9/L
* Platelet count > 50 x 10^9/L
* Hemoglobin > 8.0 g/dL without transfusion or growth factor support for at least 7 days prior to screening (with the exception of pegylated granulocyte-colony stimulating factor [G-CSF] and darbopoietin, which require at least 14 days of abstinence prior to screening)
* Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3.0 x upper limit of normal
* Estimated creatinine clearance >= 30 mL/min via Cockroft-Gault formula
* Bilirubin =< 1.5 x upper limit of normal (unless elevated bilirubin is due to Gilbert's syndrome or of non-hepatic origin)
* Prothrombin time (PT)/international normalized ratio (INR) and partial thromboplastin time (PTT) (activated partial thromboplastin time [aPTT]) =< 1.5 x upper limit of normal
* Female subjects who are of non-reproductive potential (ie, post-menopausal by history - no menses for >= 1 year; OR history of hysterectomy; OR history of bilateral tubal ligation; OR history of bilateral oophorectomy); female subjects of childbearing potential must have a negative serum pregnancy test upon screening
* Male and female subjects who agree to use both a highly effective method of birth control (eg, implants, injectables, combined oral contraceptives, some intrauterine devices [IUDs], sexual abstinence, or sterilized partner) and a barrier method (eg, condoms, vaginal ring, sponge, etc) during the period of therapy and for 30 days after the last dose of study drug for females and 90 days after the last dose of the study drug for males
* Between day +60 and day +90 after allogeneic HCT

Exclusion Criteria:

* EXCLUSION CRITERIA FOR ENROLLMENT (PRE-TRANSPLANT): Active involvement of the central nervous system with malignancy (previous central nervous system [CNS] involvement is allowed if clearance of CNS disease has been documented prior to enrollment)
* EXCLUSION CRITERIA FOR ENROLLMENT (PRE-TRANSPLANT): Pregnant or breastfeeding
* EXCLUSION CRITERIA FOR ENROLLMENT (PRE-TRANSPLANT): Karnofsky performance status < 60%
* EXCLUSION CRITERIA FOR ENROLLMENT (PRE-TRANSPLANT): Active leukemia (> 5% leukemic blasts in peripheral blood or bone marrow)
* EXCLUSION CRITERIA FOR ENROLLMENT (PRE-TRANSPLANT): Non-hematologic malignancy with a life expectancy of < 5 years
* EXCLUSION CRITERIA FOR ENROLLMENT (PRE-TRANSPLANT): Known history of human immunodeficiency virus (HIV) or active hepatitis C virus (HCV) or hepatitis B virus (HBV) infection; subjects who are positive for hepatitis B core antibody or hepatitis B surface antigen must have a negative polymerase chain reaction (PCR) result before enrollment; those who are PCR positive will be excluded
* EXCLUSION CRITERIA FOR ENROLLMENT (PRE-TRANSPLANT): Known bleeding disorders (eg, von Willebrand's disease) or hemophilia
* EXCLUSION CRITERIA FOR ENROLLMENT (PRE-TRANSPLANT): History of other malignancies, except:

  * Malignancy treated with curative intent and with no known active disease present for >= 3 years before the first dose of study drug and felt to be at low risk for recurrence by treating physician
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease Adequately treated carcinoma in situ without evidence of disease
* EXCLUSION CRITERIA (PRIOR TO IBRUTINIB ADMINISTRATION): Active and uncontrolled acute GVHD grades III or IV
* EXCLUSION CRITERIA (PRIOR TO IBRUTINIB ADMINISTRATION): Use of secondary therapy for acute GVHD at any time (defined as any systemic therapy intended to treat acute GVHD besides corticosteroids)
* EXCLUSION CRITERIA (PRIOR TO IBRUTINIB ADMINISTRATION): Requirement for anticoagulation with warfarin or other vitamin K antagonists (concomitant use of other anticoagulants is permitted)
* EXCLUSION CRITERIA (PRIOR TO IBRUTINIB ADMINISTRATION): Relapsed leukemia (> 5% leukemic blasts in peripheral blood or bone marrow after allogeneic HCT)
* EXCLUSION CRITERIA (PRIOR TO IBRUTINIB ADMINISTRATION): Karnofsky performance status < 60%
* EXCLUSION CRITERIA (PRIOR TO IBRUTINIB ADMINISTRATION): Chemotherapy =< 21 days prior to first administration of study treatment and/or monoclonal antibody =< 6 weeks prior to first administration of study treatment
* EXCLUSION CRITERIA (PRIOR TO IBRUTINIB ADMINISTRATION): Vaccinated with live, attenuated vaccines within 4 weeks of first dose of study drug
* EXCLUSION CRITERIA (PRIOR TO IBRUTINIB ADMINISTRATION): Currently active, clinically significant cardiovascular disease, such as uncontrolled arrhythmia or class 3 or 4 congestive heart failure as defined by the New York Heart Association Functional Classification; or a history of myocardial infarction, unstable angina, or acute coronary syndrome within 6 months prior to randomization
* EXCLUSION CRITERIA (PRIOR TO IBRUTINIB ADMINISTRATION): History of stroke or intracranial hemorrhage within 6 months prior to screening
* EXCLUSION CRITERIA (PRIOR TO IBRUTINIB ADMINISTRATION): Any life threatening illness, medical condition, or organ system dysfunction that, in the investigator's opinion, could compromise the subject's safety or put the study outcomes at undue risk
* EXCLUSION CRITERIA (PRIOR TO IBRUTINIB ADMINISTRATION): Major surgery within 4 weeks of first dose of study drug
* EXCLUSION CRITERIA (PRIOR TO IBRUTINIB ADMINISTRATION): Any uncontrolled active systemic infection
* EXCLUSION CRITERIA (PRIOR TO IBRUTINIB ADMINISTRATION): Unresolved toxicities from prior anti cancer therapy, defined as having not resolved to Common Terminology Criteria for Adverse Event (CTCAE, version 4), grade =< 1, or to the levels dictated in the inclusion/exclusion criteria with the exception of alopecia
* EXCLUSION CRITERIA (PRIOR TO IBRUTINIB ADMINISTRATION): Unable to swallow capsules or malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel, symptomatic inflammatory bowel disease or ulcerative colitis, or partial or complete bowel obstruction
* EXCLUSION CRITERIA (PRIOR TO IBRUTINIB ADMINISTRATION): Requires treatment with a strong cytochrome P450 (CYP) 3A4/5 inhibitor
* EXCLUSION CRITERIA (PRIOR TO IBRUTINIB ADMINISTRATION): Unwilling or unable to participate in all required study evaluations and procedures
* EXCLUSION CRITERIA (PRIOR TO IBRUTINIB ADMINISTRATION): Unable to understand the purpose and risks of the study and to provide a signed and dated informed consent form (ICF) and authorization to use protected health information (in accordance with national and local subject privacy regulations)
* EXCLUSION CRITERIA (PRIOR TO IBRUTINIB ADMINISTRATION): Currently active, clinically significant hepatic impairment (Child-Pugh class B or C)
* EXCLUSION CRITERIA (PRIOR TO IBRUTINIB ADMINISTRATION): Lactating or pregnant
* EXCLUSION CRITERIA (PRIOR TO IBRUTINIB ADMINISTRATION): Uncontrolled cardiac arrhythmias

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Rezvani, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jagasia MH, Greinix HT, Arora M, Williams KM, Wolff D, Cowen EW, Palmer J, Weisdorf D, Treister NS, Cheng GS, Kerr H, Stratton P, Duarte RF, McDonald GB, Inamoto Y, Vigorito A, Arai S, Datiles MB, Jacobsohn D, Heller T, Kitko CL, Mitchell SA, Martin PJ, Shulman H, Wu RS, Cutler CS, Vogelsang GB, Lee SJ, Pavletic SZ, Flowers ME. National Institutes of Health Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host Disease: I. The 2014 Diagnosis and Staging Working Group report. Biol Blood Marrow Transplant. 2015 Mar;21(3):389-401.e1. doi: 10.1016/j.bbmt.2014.12.001. Epub 2014 Dec 18. PMID 25529383

RESULTS

PARTICIPANT FLOW:
Groups:
- Prevention (Ibrutinib): Beginning 60-90 days after allogeneic hematopoietic cell transplantation (HCT), patients receive ibrutinib orally (PO) once daily (QD) for up to 18 months post-transplant in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Prevention (Ibrutinib)
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Prevention (Ibrutinib)
Number analyzed (Participants) | 8
Age, Customized [Count of Participants; unit: Participants]
  50-59 | 2
  60-69 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8
Diagnosis [Count of Participants; unit: Participants]
  Acute leukemia | 4
  Acute myeloid leukemia | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Relapsed Leukemia
Description: Relapsed leukemia is defined as > 5% leukemic blasts detected in bone marrow or peripheral blood. Participants were also be considered to have relapsed leukemia if they receive any active treatment for progressive leukemia after allogeneic HCT, even if they have < 5% leukemic blasts. Withdrawal of immunosuppression alone is not considered an active treatment for progressive disease.
Time Frame: Up to 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Prevention (Ibrutinib)
Number analyzed (Participants) | 8
Participants
  Relapsed | 3
  Not relapsed | 5

2. Secondary Outcome: Number of Participants With Acute Graft-versus-host Disease (GVHD) (Any Grade)
Description: Acute GVHD grades II-IV and III-IV was evaluated according to the following criteria.
  Stage of Acute GvHD was assessed as follows.
  * Stage 1: Skin: rash < 25% of skin. Liver: bilirubin 2 to 3 mg/dL. Gut: diarrhea >500 mL/day or upper-gut symptoms with positive histology
  * Stage 2: Skin: rash 25 to 50% of skin. Liver: bilirubin 3 to 6 mg/dL. Gut: diarrhea >1000 mL/day.
  * Stage 3: Skin: rash > 50% of skin. Liver: bilirubin 6 to 15 mg/dL. Gut: diarrhea > 1500 mL/day.
  * Stage 4: Skin: generalized erythroderma with bulla formation. Liver: bilirubin > 15 mg/dL. Gut: diarrhea > 2500 mL/day or severe abdominal pain with or without ileus
  Grade of Acute GvHD was determined as follows.
  * Grade 1: Stage 1-2 Skin + No Liver stage + No Gut stage
  * Grade 2: Stage 3 Skin OR Stage 1 Liver or Stage 1 Gut
  * Grade 3: No Skin stage + Stage 2 to 3 Liver Stage 2 to 4 Gut
  * Grade 4: Stage 4 Skin + or Stage 2 to 3 Liver + No Gut stage
Time Frame: At 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | Prevention (Ibrutinib)
Number analyzed (Participants) | 8
Participants | 4

3. Secondary Outcome: Number of Participants With Chronic GVHD
Description: Assessment of chronic GvHD was performed using the 2015 NIH consensus criteria.
Time Frame: At 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Prevention (Ibrutinib)
Number analyzed (Participants) | 8
Participants | 3

4. Secondary Outcome: Number of Participants Negative for Detectable Minimal Residual Disease
Description: Detectable minimal residual disease was assessed using high-throughput sequencing (ClonoSEQ) and high-sensitivity flow cytometry. Minimal residual disease was considered present if > 1 x 10^-6 leukemic clones are detected by ClonoSEQ, or if any aberrant blasts matching the original leukemic immunophenotype are detected by high-sensitivity flow cytometry.
Time Frame: day +90, day +180, 1 year, 1.5 years
Population: Participants who had minimal residual disease testing at the respective time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Prevention (Ibrutinib)
Number analyzed (Participants) | 8
Participants
  day +90 | 8
  day +180: number analyzed (Participants) | 7
  day +180 | 7
  1 year: number analyzed (Participants) | 5
  1 year | 5
  1.5 years: number analyzed (Participants) | 5
  1.5 years | 5

ADVERSE EVENTS:
Time Frame: up to 18 months
Arm/Group | Prevention (Ibrutinib)
All-Cause Mortality (participants affected / at risk) | 2/8
Serious Adverse Events (participants affected / at risk) | 3/8
Other Adverse Events (participants affected / at risk) | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prevention (Ibrutinib) (N=8)
Pancytopenia (Blood and lymphatic system disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Fever (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prevention (Ibrutinib) (N=8)
Anorexia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Peripheral Neuropathy (Nervous system disorders) | 1
Leg Pain (Musculoskeletal and connective tissue disorders) | 1
Bilateral Hand Pain (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Shortness of breath (dyspnea) (Respiratory, thoracic and mediastinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Abdominal Pain (Gastrointestinal disorders) | 1
Oral Ulcer (Gastrointestinal disorders) | 1
Facial hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 1
Itchy Skin (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
Blepharitis (Eye disorders) | 1
Imbalance (General disorders) | 1
Edema, bilateral (General disorders) | 1

LIMITATIONS AND CAVEATS:
This study did not enroll the planned number of participants and did not achieve statistical power.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-23): https://cdn.clinicaltrials.gov/large-docs/86/NCT03267186/Prot_SAP_001.pdf
  • Informed Consent Form (2020-12-08): https://cdn.clinicaltrials.gov/large-docs/86/NCT03267186/ICF_000.pdf